CLINICAL TRIAL: NCT06031779
Title: Application of Serum Bile Acid Profile in the Diagnosis of Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Principal Investigator,Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20232258-C-1
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer
Keywords: serum bile acid; biomarker
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- gastric cancer
- non-gastric cancer

SUMMARY:
In this study, the composition and level of serum bile acids in patients with gastric cancer and non-gastric cancer were analyzed by detecting the serum bile acid profile, so as to develop new serological diagnostic methods for early diagnosis and treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-70, both gender;
2. The gastric cancer group was early gastric cancer or advanced gastric cancer diagnosed by endoscopic examination and pathological biopsy. The non-gastric cancer group included patients without gastric lesions, superficial gastritis, chronic atrophic gastritis, intestinal metaplasia or dysplasia diagnosed by gastroscopy or pathological biopsy;
3. Informed consent was obtained.

Exclusion Criteria:

1. The patients have diseases that affect bile acid metabolism, such as liver cirrhosis, gallstones or inflammatory bowel disease, Behcet's disease, etc;
2. Due to other diseases, the patient took drugs affecting bile acid metabolism, such as cholestyramine, anti-inflammatory Lidan tablets, Danshu capsules, ursodeoxycholic acid, obticholic acid, Schisandrin B, tanshinone ⅡA, Yinzhihuang, etc;
3. Pregnant women;
4. Primary tumors of other systems were diagnosed;
5. Those with poor physiopathological conditions, such as chronic kidney disease requiring long-term dialysis;
6. Patients with mental illness;
7. Patients who have received radiotherapy or surgery previously;
8. Those with poor adherence or difficult to follow up.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending Xijing Hospital and Patients included in the biospecimen bank
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
serum bile acid profile before treatment | 1 month

SECONDARY OUTCOMES:
concentration of serum tumor markers before treatment | 1 month
  CEA, CA19-9 and CA12-5

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Shi, PhD, Study Director — Xijing Hpsipital of Digestive Disease
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China